CLINICAL TRIAL: NCT06277778
Title: Effect of Combined Music and Taekwondo Training on the Psychological and Physical Condition of Children with Autism Spectrum Disorder: a Randomized Controlled Trial
Brief Title: Effect of Combined Music and Taekwondo Training for Children with Autism Spectrum Disorder
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20211117003-03
Record Dates: First submitted 2024-01-14; First posted 2024-02-26 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Autism Spectrum Disorder
Keywords: music; taekwondo; Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Taekwondo training with music therapy (Experimental): the participating children will attend 20 sessions of Taekwondo training with the presence of music.
  Interventions: Other: Taekwondo training with music therapy
- Taekwondo training alone (Sham Comparator): the participating children will attend 20 sessions of Taekwondo training alone.
  Interventions: Other: Taekwondo training alone

INTERVENTIONS:
Other: Taekwondo training with music therapy — Taekwondo training with music therapy
  Arms: Taekwondo training with music therapy
Other: Taekwondo training alone — Taekwondo training without music therapy
  Arms: Taekwondo training alone

SUMMARY:
The goal of this randomized controlled trial is to evaluate the effect of combined music and taekwondo training on the mental and physical condition of children with autism spectrum disorder. Participants will be asked to do combined music and taekwondo training or taekwondo training alone to evaluate if the combined training is better than the taekwondo training alone on mental and physical performance for children with autism spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

* Chinese children aged 7 to 9 years who have been clinically diagnosed as ASD by developmental paediatricians or clinical psychologists based on the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition criteria for ASD.

Exclusion Criteria:

* children who have experience in Taekwondo training;
* children who have received music therapy within the previous 12 months;
* those who have severe sensory disorders (blindness or deafness);
* those who have underlying congenital abnormalities or other diseases that limit their ability to engage in physical activities.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-06-30 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Engagement in the Training Sessions | Through training completion, an average of 20 sessions over 10 consecutive weeks
  the Revised Individual Child Engagement Record (ICER); The ICER-R uses a 15-second momentary time sampling approach and involves the coding of types of engagement, the occurrence of interaction and the interaction partner (coach or peers), and whether the child was physically prompted. The types of engagement being coded at each 15-second interval are active engagement, passive engagement, active non-engagement, and passive non-engagement.
Gross Motor Skills | Baseline, 10 weeks
  Motor skills will be assessed using the Bruininks-Oseretsky Test of Motor Proficiency-2

SECONDARY OUTCOMES:
Physical Activity Level | Through training completion, an average of 20 sessions over 10 consecutive weeks
  Participants will wear an optical heart rate monitor on their forearm to measure their exercise heart rate as a reflection of the physical activity level during the training. Continuous heart rate data will be recorded for every record and expressed as the mean heart rate per min.
Enjoyment State | Through training completion, an average of 20 sessions over 10 consecutive weeks
  The Children's Emotional Manifestation Scale (CEMS) will be used to assess the children's emotional state. It classifies observable emotional behaviours into five categories: 'Facial expression', 'Vocalization', 'Activity', 'Interaction', and 'Level of cooperation'. Each category is scored from 1 to 5. The numbers obtained for each category are added together to obtain the total score, which will be between 5 and 25. High scores indicate the manifestation of more negative emotional behavior.
Rate of Perceived Exertion | Through training completion, an average of 20 sessions over 10 consecutive weeks
  Children will be asked to rate their exertion level using the Borg 6-to-20 Scale, in which "6" indicates "no exertion at all" and "20" indicates "maximal exertion".
Taekwondo skills performance | Baseline, 10 weeks
  A scoring system was modified for use in this project with reference to the international Taekwondo referee scoring standard. Children's performance for a set of selected Taekwondo moves and kicks will be observed and scored by two qualified referees. The performance will be scored out of 8 marks, with 3 marks for presentation, 2 marks for cognitive ability, 2 marks for basic skills, and 1 mark for social interaction. Higher scores indicate better performance.
Conners' Continuous Performance Test II | Baseline, 10 weeks
  This test will be used to measure the children's selective attention, that is, their ability to maintain a consistent focus on some continuous stimuli.
Comprehensive Trail-Making Test (CTMT) | Baseline, 10 weeks
  The test consists of five visual search and sequencing tasks that are heavily influenced by attention, concentration, resistance to distraction, and cognitive flexibility (or set-shifting). The child is required to connect a series of stimuli (numbers, expressed as numerals or in word form, and letters) in a specified order as fast as possible in each trial. The time scores for the five CTMT trials will be converted to standardized T-scores according to the reference tables in the testing manual, and be summed up to produce a global performance level score, the CTMT Composite Index (CI), which can then be converted into a percentile score according to the participant's chronological age. Higher T score and CTMT CI correspond to better performance.
Social Responsiveness Scale, second edition (SRS-2) | Baseline, 10 weeks
  This scale will be completed by the parents. It is a 65-item autism rating scale widely use to identify a spectrum of deficits in reciprocal social behavior, ranging from absent to severe, based on observations of a child's behavior in various social settings. Scoring is on a four-point Likert Scale with five subscales (social awareness, social cognition, social communication, social motivation, and autistic mannerism). Higher T-scores correspond to poorer social functioning.
Childhood Autism Spectrum Test | Baseline, 10 weeks
  This is a 39-item, yes-or-no questionnaire of children's social behavior and communication tendencies as reported by their parents. The questionnaire has been translated into Chinese and is being validated. The cut-off score of 15 marks indicates possible autism spectrum disorder (ASD) or related social-communication difficulties.
Strength and Difficulties Questionnaires (SDQ) | Baseline, 10 weeks
  The questionnaire will be completed by parents. There are 25 items in the SDQ, which consists of five scales, each with five items, for assessing children's mental health status in terms of emotional, conduct, hyperactivity, peer problems, and prosocial behavior.
Clinical Global Improvement (CGI) score | 10 weeks, 2 months follow-up
  The CGI-I will be completed by parents to evaluate children's functional changes in daily life after completion of the 10-week program, and at 2-month follow-up. The CGI-I consisted of 12 questions developed by our research team, which are focused on all core symptoms of ASD and covered the following aspects: (1) motor functioning; (2) children's capability to follow instructions; (3) social, communication, and language understanding and expression; and (4) children's capabilities for attention shifting, attention to complete a task, attention to details, and imagination.

CONTACTS AND LOCATIONS:
Overall Officials: Clare CW YU, PhD, Principal Investigator — Assistant Professor
Locations (1):
- Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yu CCW, Mok KM, Mak E, Au CT, Chan DFY, Wu S, Chung RCK, Ip MCK, Wong SWL. Protocol for evaluating the effects of integrating music with taekwondo training in children with autism spectrum disorder: A randomized controlled trial. PLoS One. 2025 Jan 31;20(1):e0315503. doi: 10.1371/journal.pone.0315503. eCollection 2025. PMID 39888930